CLINICAL TRIAL: NCT06109454
Title: Observational Study on the Efficacy and Safety of Huaier Granules Compared With Platinum Containing Dual Drug Combination Chemotherapy in Adjuvant Therapy for Resectable Stage II-IIIA Non-small Cell Lung Cancer After Radical Surgery
Brief Title: Observation on the Therapeutic Effect of Huaier Granules in the Adjuvant Treatment of Non-small Cell Lung Cancer After Radical Surgery
Status: Recruiting | Type: Observational
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry); Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hongxu Liu, professor, Liaoning Cancer Hospital & Institute
Other Study IDs: HE-202306
Record Dates: First submitted 2023-10-24; First posted 2023-10-31 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Huaier granule; Non-small Cell Lung Cancer; Efficacy; Safety
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Huaier Granule: The subjects voluntarily gave up postoperative adjuvant therapy, including chemotherapy, targeted therapy, immunotherapy, and radiation therapy, and agreed to take Huaier granules.
  Interventions: Drug: Huaier granule
- Control: The subjects received standard platinum dual-drug chemotherapy.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Huaier granule — The subjects voluntarily gave up postoperative adjuvant therapy, including chemotherapy, targeted therapy, immunotherapy, and radiation therapy, and agreed to take Huaier granules.The subjects took Huaier granules orally, one bag (10g) per time, three times a day. Until the end of the study, intolerable toxicity, withdrawal from the study for any reason or death, or when the researcher determines that there is no further benefit, whichever occurs first. Please refer to the drug manual for specific usage. It is recommended that patients start taking Huaier granules 1-2 weeks after surgery.
  Other Names: Z20000109（NMPA Approval Number）
  Groups: Huaier Granule
Other: Control — The subjects received standard platinum dual drug chemotherapy.The subjects were treated with carboplatin injection (300mg/m2, intravenous injection, first day) combined with pemetrexed disodium (pathological type: adenocarcinoma, intravenous injection, 500mg/m2) or albumin bound paclitaxel (pathological type: squamous cell carcinoma, 260mg/m2, intravenous injection, first day) every three weeks, with a maximum of four cycles.
  Groups: Control

SUMMARY:
This study is a multicenter, prospective, and observational clinical study aimed at exploring whether the 3-year DFS in the Huaier group is not inferior to the control group receiving standard platinum dual-drug chemotherapy.

DETAILED DESCRIPTION:
This study is a small sample observational study, mainly exploring whether the 3-year DFS of the Huaier group is not inferior to the control group receiving standard platinum dual drug chemotherapy. Therefore, this study will conduct a small sample exploratory analysis. It is expected to include 240 non-small cell lung cancer patients who have been diagnosed with stage Ⅱ-ⅢA and are eligible for surgery at selected research centers from April 2023 to July 2025. Among them, 120 patients in the Huaier Granule group refused to undergo adjuvant chemotherapy due to reasons such as intolerance or disagreement, and agreed to receive Huaier Granule monotherapy as an adjuvant treatment; There are 120 patients in the control group, all of whom plan to receive standard chemotherapy as an adjuvant treatment plan (including platinum based dual-drug combination chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age ≤ 75, regardless of gender.
* Confirmed as non-small cell lung cancer by histopathology, with pathological staging of stage Ⅱ-ⅢA.
* Received radical R0 resection of lung cancer within 2 months before enrollment, and did not receive any postoperative adjuvant therapy or preoperative neoadjuvant therapy.
* ECOG（Eastern Cooperative Oncology Group）score:0-2.
* The patient voluntarily participated in the study, agreed to cooperate with the researcher for data collection, and signed an informed consent form.

Exclusion Criteria:

* Known to be allergic to the components of Huaier granules or avoid or use Huaier granules with caution (Huaier group).
* Those who have difficulty swallowing, complete or incomplete gastrointestinal obstruction, active gastrointestinal bleeding, perforation, and other causes of difficulty in taking oral medication.
* Non-small cell lung cancer patients who plan to receive targeted therapy, immunotherapy, chemotherapy combined with immunotherapy, radiotherapy, synchronous radiotherapy and chemotherapy during the study period.
* The patient has a history of other new malignant tumors within 5 years.
* The expected survival time of the patient is less than half a year.
* Surgical complications that have not recovered or are accompanied by severe infections after radical resection of lung cancer.
* Pregnant or lactating women or planned pregnancy preparation.
* The patient has received other traditional Chinese patent medicines and simple preparations with anti-tumor effect in the past one month (including but not limited to compound cantharidin capsule, cinobufagin capsule, Kangai injection, Brucea javanica injection, etc., the specific instructions shall prevail).
* The patient suffers from severe mental illness or other reasons that the researcher deems unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is resectable stage Ⅱ-ⅢA non-small cell lung cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival (DFS) rate | start of treatment until 3-year follow-up
  The proportion of participants who did not experience disease recurrence or death within 3 years after undergoing lung cancer radical surgery.

SECONDARY OUTCOMES:
1-year or 2-year DFS rate | start of treatment until 1-year or 2-year follow-up
  The proportion of participants who did not experience disease recurrence or death within 1 or 2 years after undergoing lung cancer radical surgery
1-year, 2-year or 3-year overall survival (OS) rate | start of treatment until 1-year, 2-year or 3-year follow-up
  The proportion of subjects who survived within 1 year, 2 years or 3 years after undergoing radical lung cancer surgery among all subjects.
1-year, 2-year or 3-year local recurrence free survival (LRFS) rates | start of treatment until 1-year, 2-year or 3-year follow-up
  The proportion of subjects who did not experience local recurrence of lung cancer within 1 year, 2 years or 3 years after undergoing radical lung cancer surgery.
1-year, 2-year or 3-year distant metastasis free survival (DMFS) rates | start of treatment until 1-year, 2-year or 3-year follow-up
  The proportion of subjects who did not experience distant metastasis within 1 year, 2 years, or 3 years after undergoing lung cancer radical surgery
Quality of Life Score (SF-36 Scale) | start of treatment until 3-year follow-up
  The Health Survey Short Form[(SF-36 Scale (Chinese Version) ]developed by the US Medical Bureau research team was used for evaluation. The scale has 36 items and aims to evaluate the health and functional status of multiple age groups, different diseases, and control populations.Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
The incidence and severity of adverse events (AE) and severe adverse events (SAE) | start of treatment until 3-year follow-up
  The definitions and severity grading of AE and SAE can refer to the corresponding descriptions in the definition and evaluation section of AE. The incidence rate is defined as the proportion of subjects who have experienced AE and SAE to the corresponding total population.

OTHER OUTCOMES:
Changes in peripheral blood lymphocyte subpopulations | start of treatment until 3-year follow-up
  Observe and describe the changes in peripheral blood lymphocyte subpopulations from baseline, peripheral blood lymphocyte subpopulations include but are not limited to CD3+T, CD4+T, and CD8+T.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxu Liu, PhD, Principal Investigator — Liaoning Cancer Hospital & Institute
Locations (1):
- Liaoning Cancer Hospital & Institute, Shenyang, Liaoning, China